CLINICAL TRIAL: NCT04461574
Title: Clinical Trial Comparing the Use of Orcellex® Brush Versus Cervex-Brush® on Vaginal Vault Smear Cytology Adequacy Rate in Patients Treated With Radiotherapy for Cervical Cancer
Brief Title: Orcellex® Brush Versus Cervex-Brush® on Vault Smear Adequacy in Patients Treated With Radiotherapy for Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, He Mung Yuen, Associate Consultant, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 147-06
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervex Brush (Placebo Comparator)
  Interventions: Device: Orcellex Brush
- Orcellex Brush (Active Comparator)
  Interventions: Device: Cervex Brush

INTERVENTIONS:
Device: Orcellex Brush — Subjects will receive vaginal vault smear using both Orcellex Brush and Cervex Brush at the same follow-up visit, with order of smear taking decided by randomization.
  Arms: Cervex Brush
Device: Cervex Brush — Subjects will receive vaginal vault smear using both Orcellex Brush and Cervex Brush at the same follow-up visit, with order of smear taking decided by randomization.
  Arms: Orcellex Brush

SUMMARY:
Vaginal vault cytology is commonly used for follow-up surveillance in patients treated for cervical cancer. It is known that the smear inadequacy rate is high, especially in patients post-radiotherapy at 10%. The current practice is to use Cervex-Brush®, which was designed for cervical smear taking. Cervix will shrink into a dimple with a flat vaginal vault and vagina may be stenotic after radiotherapy, rendering the use of the conventional sampling device difficult. Orcellex® Brush was designed to collect cells from oral mucosa, with high patient satisfaction and low smear inadequacy of 1% in one study. As both the vaginal vault mucosa and oral mucosa are flat surface lined with stratified squamous epithelium, the use of Orcellex® Brush in vaginal vault smear appeared applicable. It has a smaller head with a flat surface of hair, which might better fit the flat vault surface and narrow vaginal canal. It is postulated that the Orcellex® Brush helps in improving vaginal vault smear adequacy rate in patients after radiotherapy treatment for cervical cancer.

DETAILED DESCRIPTION:
Patients with cervical cancer treated with primary irradiation will be recruited at their routine post-treatment surveillance follow-up in the out-patient clinic, in the order of their appointment time. Study procedure will be explained and written informed consent is obtained from each subject at the visit. Systemic and vaginal examination will be carried out as usual. Subjects will receive vaginal vault smear by both Cervex-Brush® and Orcellex® Brush during the same speculum examination. The order of using smear sampling devices will be randomized. Randomization will be carried out according to computer-generated random numbers, allocated by sequentially numbered, sealed opaque envelopes. Subjects will be randomized into two groups: using Cervex-Brush® first followed by Orcellex® Brush, or vice versa. The procedure of smear taking will be carried out by four trained clinicians who are independent of the study. The method of smear taking will be standardized for both Cervex-Brush® and Orcellex® Brush. The vaginal vault will be swept horizontally by the brush and the cervical dimple, if seen, will be rotated five times by the brush. Each sampling device will be shaken vigorously in separate Thinprep specimen containers, which is labelled as smear A for Cervex-Brush® and smear B for Orcellex® Brush.

The subjects are unaware of the sequence of the sampling device used, as they cannot see the procedure of smear taking during examination. The patient will be asked about the pain score during each smear taking, by using the visual analog scale. Any vaginal bleeding will be recorded.

The specimen will be sent to the laboratory and will be processed by the ThinPrep method. The cytopathologist is unaware as to which device is used for that particular specimen and the slide prepared from it. One pathologist will be responsible in screening all the vault smears involved in this study. Adequacy of vault smear sample was defined by the Bethesda System as a minimum of 2000 well-visualized and well-preserved squamous cells.

Patients will be arranged subsequent follow-up visits at appropriate time interval according to the department protocol. Patients with inadequate smear result by both sampling devices will be called back early within 8 weeks for repeat smear using the conventional Cervex-Brush®.

Patients with cervical cancer in the department will have surveillance follow-ups at variable intervals from 3 months to 12 months, depending on the time interval from previous treatment and patients' symptoms. Some patients may have repeated smears during the study period. As the result of previous smear will have no impact on the adequacy rate of subsequent smear, patients can be recruited for smear taking more than once in the study. Hence the actual number of patients recruited in the study would be less than the calculated sample size of 160.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical cancer treated with primary radiotherapy
* Patients aged 18 years or older
* Patients requiring vaginal vault cytology for follow-up surveillance

Exclusion Criteria:

* Patients who refuse vaginal examination or vaginal vault smear at follow-up.
* Patients who have visible tumour at vaginal vault requiring direct biopsy at speculum examination.
* Patients who cannot understand the study purpose and procedure.
* Patients who cannot read the words written in Chinese or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Vault cytology adequacy rate | through study completion, an average of 1 year
  Adequacy of vault smear sample was defined by the Bethesda System as a minimum of 2000 well-visualized and well-preserved squamous cells

SECONDARY OUTCOMES:
Patient pain score | through study completion, an average of 1 year
  Pain score 0-10 by visual analog scale higher score means higher level of pain minimum = 0 maximum = 10
Vaginal bleeding | through study completion, an average of 1 year
  Any bleeding noted by investigators during per vaginal examination
Detection of abnormal cytology | through study completion, an average of 1 year
  Any detection of abnormal cells by vault cytology
borderline cellularity rate | through study completion, an average of 1 year
  borderline cellularity requiring further clarification

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] So YL, He MY, Hui SK, Yu EL. Clinical trial comparing the use of Orcellex(R) Brush versus Cervex-Brush(R) on vaginal vault smear cytology adequacy rate in patients treated with radiotherapy for cervical cancer. J Gynecol Oncol. 2025 May;36(3):e43. doi: 10.3802/jgo.2025.36.e43. Epub 2024 Oct 22. PMID 39453394